CLINICAL TRIAL: NCT01869283
Title: Effectiveness of Physical Therapy Treatments of Myofascial Trigger Points in Subjects With Neck Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Rinaldo Roberto de Jesus Guirro, Professor, PT, PhD, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: U1111-1143-4456
Record Dates: First submitted 2013-05-27; First posted 2013-06-05 (Estimated); Last update posted 2013-06-05 (Estimated); Status verified 2013-05

CONDITIONS: Neck Pain; Myofascial Pain Syndrome
Keywords: Physical Therapy Modalities; Myofascial Pain Syndromes; Skeletal Muscle
MeSH Terms: conditions — Neck Pain; Myofascial Pain Syndromes | interventions — High-Energy Shock Waves

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Kinesiotherapy group (Experimental): The volunteer will be subjected to the following protocol: cervical traction, 3 sets of 1 minute, 30-second rest between sets; mobilization grade III postero-anterior on the spines processes of vertebrae C2 to C7, 10 oscillations for each vertebrae; myofascial release of the upper trapezius muscle, 3 sets of 1 minute for each side; static stretching of the upper trapezius muscle, 3 sets of 30 seconds, with an interval of 10 seconds between sets.
  Interventions: Other: Kinesiotherapy
- kinesiotherapy + static ultrasound group (Experimental): Same protocol group kinesiotherapy + ultrasound on the trigger points of the upper trapezius muscle in a static way, with 1 MHz, continuous dose of 1.5 W/cm2, for 1.5 minutes.
  Interventions: Other: Kinesiotherapy; Other: Ultrasound
- kinesiotherapy + diadynamic currents group (Experimental): Same protocol group kinesiotherapy + diadynamic currents, with negative electrode (7.0 x 7.0 cm) placed on the myofascial trigger point, while the positive electrode (7.0 x 7.0 cm) is placed between the shoulder blades. Will apply 4 minutes from the biphasic mode (DF) and 6-minute short period (CP), the first of which intesidade the sensory threshold and the second threshold motor, both bearable for the patient.
  Interventions: Other: Kinesiotherapy; Other: Diadynamic currents
- Control group (No Intervention): The volunteers of this group will not be subjected to any form of treatment, was evaluated in three stages, as the other groups. It is noteworthy that, after the volunteer's participation, will be offered at the same physical therapy for myofascial pain.

INTERVENTIONS:
Other: Kinesiotherapy
  Arms: Kinesiotherapy group; kinesiotherapy + diadynamic currents group; kinesiotherapy + static ultrasound group
Other: Ultrasound
  Arms: kinesiotherapy + static ultrasound group
Other: Diadynamic currents
  Arms: kinesiotherapy + diadynamic currents group

SUMMARY:
Neck pain is a prevalent musculoskeletal dysfunction. Studies point that individuals with chronic pain have metabolic, vascular and electromyographic changes in trapezius muscle. Moreover, a common clinical sign in this muscle in subjects with neck pain is the presence of myofascial trigger points. These are related to the sensory, motor and autonomic changes, being defined as palpable nodules located in the taut band of skeletal muscle. In this context, the focus on treatment modalities stands out in the literature, however, other resources commonly used in clinical practice still lack scientific evidence. Therefore, the aim of this project is to evaluate the effectiveness of physiotherapy resources in the treatment of myofascial trigger points in the trapezius muscle of patients with neck pain. For such, volunteers with neck pain for more than 90 days, of both genders, aged between 18 and 59 years and bilateral myofascial trigger points in the upper trapezius will be randomized into the following groups: group 1 (kinesiotherapy, n = 20), group 2 (kinesiotherapy + static ultrasound, n = 20), group 3 (kinesiotherapy + diadynamic currents, n = 20) and group 4 (untreated control, n = 20). Volunteers will undergo ten sessions of treatment, being realized the following evaluations: surface electromyography, infrared thermography, numerical scale of pain assessment, algometry, Neck Disability Index and skin impedance. For data analysis, normality test will used to verify the data distribution and consistent statistical test for the appropriate comparisons within and between groups, and thus considered two factors in the comparisons, time and group. Will adopt a significance level of 5%.

ELIGIBILITY:
Inclusion Criteria:

* neck pain for more than 90 days
* aged 18 to 59 years
* presence of trigger points in the upper trapezius muscle

Exclusion Criteria:

* history of trauma to the neck
* surgery in the head, face or neck
* herniated cervical
* degenerative diseases of the spine
* systemic diseases
* underwent physical therapy in the last three months
* analgesics, anti-inflammatories or muscle relaxants last week
* medical diagnosis of fibromyalgia
* body mass index (BMI) greater than 28 kg/m2
* signs and symptoms of depression

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2013-05; Primary Completion 2016-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Pain | 3 years
  Will be apply the following assessment tools: Neck Disability Index (assesses neck pain and disability), algometry (evaluates pressure pain threshold), and numerical scale of pain assessment (assesses pain intensity).

SECONDARY OUTCOMES:
Cervical range of motion | 3 years
  Through a fleximeter will be evaluated movements of flexion, extension, rotation and inclination of the neck.
Skin temperature | 3 years
  Through of thermograph will be evaluated skin temperature on myofascial trigger points.
Muscle activity | 3 years
  Through surface electromyography will be evaluated the electrical activity of the upper trapezius muscle.

CONTACTS AND LOCATIONS:
Overall Officials: Rinaldo Guirro, PhD, Principal Investigator — University of Sao Paulo
Locations (1):
- University of Sao Paulo, Ribeirão Preto, São Paulo, Brazil

REFERENCES:
- See also: Related Info — http://www.fmrp.usp.br